CLINICAL TRIAL: NCT01038661
Title: Randomized, Controlled Study Comparing the Efficacy and Safety of Docetaxel （60mg/m2）Maintenance Treatment vs. Best Supportive Care Following First Line Chemotherapy With Different Doses of Docetaxel（75/60mg/m2）in Combination With Cisplatin in Patients With Local Advanced or Metastatic （Stage IIIB/IV）Non-Small Cell Lung Cancer
Brief Title: Tax First-line Chemotherapy With Different Doses and Then Maintenance Therapy
Acronym: TFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DOCET_L_04827
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2014-02-28 (Estimated); Status verified 2014-02

CONDITIONS: Lung Neoplasms
MeSH Terms: conditions — Lung Neoplasms | interventions — Docetaxel; Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- First line treatment: docetaxel 75 mg/m² + cisplatin 75 mg/m² (Experimental): Docetaxel 75 mg/m² + cisplatin 75 mg/m² on day 1, repeated every 3 weeks, up to 4 cycles
  Interventions: Drug: Docetaxel; Drug: Cisplatin
- First line treatment:: docetaxel 60 mg/m² + cisplatin 75 mg/m² (Experimental): Docetaxel 60 mg/m² + cisplatin 75 mg/m² on day 1, repeated every 3 weeks, up to 4 cycles
  Interventions: Drug: Docetaxel; Drug: Cisplatin
- Maintenance treatment: docetaxel (60 mg/m2) (Experimental): Docetaxel 60 mg/m² on day 1, repeated every 3 weeks until progressive disease or up to 6 cycles
  Interventions: Drug: Docetaxel
- Maintenance treatment: best supportive care (BSC) (Active Comparator): BSC until progressive disease
  Interventions: Other: Best supportive care (BSC)

INTERVENTIONS:
Drug: Docetaxel — Formulation: concentrated solution for intravenous infusion (IV)
  Route(s) of administration: 1-hour IV
  Other Names: Taxotere®
  Arms: First line treatment: docetaxel 75 mg/m² + cisplatin 75 mg/m²; First line treatment:: docetaxel 60 mg/m² + cisplatin 75 mg/m²; Maintenance treatment: docetaxel (60 mg/m2)
Drug: Cisplatin — Formulation: concentrated solution for intravenous infusion (IV)
  Route(s) of administration: 1-3-hour IV
  Arms: First line treatment: docetaxel 75 mg/m² + cisplatin 75 mg/m²; First line treatment:: docetaxel 60 mg/m² + cisplatin 75 mg/m²
Other: Best supportive care (BSC) — Any treatment including palliative radiotherapy for pain relief-but not chemotherapy - that is considered appropriate by the investigator
  Arms: Maintenance treatment: best supportive care (BSC)

SUMMARY:
The Primary Objective is to evaluate the progression-free survival (PFS).

The secondary objectives are:

* To compare the disease control rates of different doses of Docetaxel+Cisplatin as first-line treatment according to Response Evaluation Criteria In Solid Tumors (RECIST) criteria;
* To evaluate the overall response rate (ORR);
* To evaluate the time to disease progression (TTP);
* To evaluate the overall survival (OS);
* To evaluate the toxicity.

DETAILED DESCRIPTION:
The study consists in:

* A first line treatment phase: participants receive 4 cycles of chemotherapy (each cycle contains 3 weeks) with either docetaxel (75 mg/m2) plus cisplatin (75 mg/m2) or docetaxel (60 mg/m2) plus cisplatin (75 mg/m2) ,
* A maintenance treatment phase: participants with disease control (complete response [CR], partial response [PR] or stable disease [SD]) after the initial treatment receive up to 6 cycles of chemotherapy with docetaxel (60 mg/m2) or best supportive care (BSC).
* A follow-up period from the end of study treatment until participant death or end of study.

ELIGIBILITY:
Inclusion criteria:

* Histologic or cytologic diagnosis of advanced non-small-cell lung cancer (NSCLC)
* Based on International Association for the Study of Lung Cancer (IASLC) 2009 new Tumor-Node-Metastasis (TNM) stage criteria of lung cancer, local advanced stage IIIB (not applicable for radical radiation therapy) disease or metastatic stage IV disease or recurrent disease
* At least one evaluable tumor lesion based on RECIST criteria (>= 20 mm with conventional techniques or >= 10 mm with spiral Computed Tomography scan)
* Eastern Cooperative Oncology Group performance status (ECOG PS) 0/1
* Adequate bone marrow reserve

  * absolute neutrophil count >= 2.0×10^9/L
  * platelets >= 100×10^9/L
  * hemoglobin >= 9.0 g/dL
* Adequate hepatic function

  * total bilirubin <= Upper Normal Limit (UNL)
  * Aspartate Amino Transferase (AST), Alanine Amino Transferase (ALT) <= 2.5 UNL
  * alkaline phosphatase (ALP) <= 5 UNL
* Adequate renal function (serum creatinine <= UNL or creatinine clearance >= 60 mL/min)
* No prior chemotherapy was allowed or only (neo) adjuvant chemotherapy ended more than 6 months before treatment (patients should not have been heavily pre-treated, the maximum cumulative dose of cisplatin allowed is 350 mg/m²)
* Prior surgery was permitted only if the operation performed more than 4 weeks ago and the patient was completely recovery
* Childbearing potential either terminated or attenuated by the use of an approved contraceptive method
* Inform consent signed

Exclusion criteria:

* Other tumour type than advanced / metastatic NSCLC in recent 5 years (except cone-biopsied carcinoma-in-situ of the cervix or adequately treated basal or squamous cell carcinoma of the skin).
* Presence of symptomatic central nervous system metastases
* Inadequate liver function

  * total bilirubin > 1 UNL
  * ALT and/or AST>1.5 UNL associated with alkaline phosphatase > 2.5 UNL
  * inadequate renal function (creatinine > 1.0 times UNL and in case of limit value, creatinine clearance < 60 mL/min)
* Prior radiation therapy, or surgery operation within 4 weeks
* Prior use of taxoids
* Active infection, or serious concomitant systemic disorder incompatible with the study
* Childbearing potential but unwilling to use of an approved contraceptive method
* Receive treatment from other clinical trials during this study treatment
* History of hypersensitivity to any of study medication
* Other serious concomitant abnormal or illness

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2009-11; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) during the maintenance treatment phase | From 2nd randomization to progression or death of any cause (every 2 cycles (6 weeks) during study treatment, and then every 8 weeks during follow-up period)

SECONDARY OUTCOMES:
Disease control rate (DCR) during the first line treatment phase | Every 2 cycles (6 weeks)
Overall response rate (ORR) during the first line treatment phase | Every 2 cycles (6 weeks)
Time to disease progression (TTP) during the maintenance treatment phase | From 2nd randomization up to disease progression (every 2 cycles (6 weeks))
Overall survival (OS) | From 1st randomization to death of any cause (every 2 cycles (6 weeks) during study treatment, and then every 8 weeks during follow-up period)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi-Aventis Administrative Office, Shanghai, China

REFERENCES:
- [Derived] Zhang L, Lu S, Cheng Y, Hu Z, Wu YL, Chen Z, Chen G, Liu X, Yang J, Zhang L, Chen J, Huang M, Tao M, Cheng G, Huang C, Zhou C, Zhang W, Zhao H, Sun Y. Docetaxel maintenance therapy versus best supportive care after first-line chemotherapy with different dose docetaxel plus cisplatin for advanced non-small cell lung cancer (TFINE study, CTONG-0904): an open-label, randomized, phase III trial. Ann Transl Med. 2021 Feb;9(4):338. doi: 10.21037/atm-20-8078. PMID 33708965